CLINICAL TRIAL: NCT02189967
Title: Postoperative Radiotherapy of Non-small Cell Lung Cancer: Accelerated vs. Conventional Fractionation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Consortium for Translational Cancer Research (Other); National Center for Radiation Research in Oncology Dresden/Heidelberg (Other); Radiation Oncology Working Group of the German Cancer Society (Other)
Responsible Party: Principal Investigator, Dr. Rebecca Bütof, Principal Investigator, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR-PORTAF-2014
Record Dates: First submitted 2014-05-22; First posted 2014-07-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; radiotherapy; accelerated fractionation; conventional fractionation; postoperative
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional fractionation (Active Comparator): radiotherapy with conventional fractionation (5 x 2Gy per week)
  Interventions: Radiation: conventional fractionation
- accelerated fraction (Active Comparator): radiotherapy with accelerated fraction (7 x 2 Gy per week)
  Interventions: Radiation: accelerated fraction

INTERVENTIONS:
Radiation: conventional fractionation — In this treatment arm patients will receive radiotherapy with the currently used conventional fractionation schedule i.e. 5 fractions per week, 2 Gy single dose.
  Arms: conventional fractionation
Radiation: accelerated fraction — In this treatment arm patients will receive radiotherapy with an accelerated fractionation schedule i.e. 7 fractions per week, 2 Gy single dose.
  Arms: accelerated fraction

SUMMARY:
In this randomized multicentric phase II study it will be investigated whether an accelerated postoperative radiotherapy with photons or protons (7 fractions per week, 2 Gy single dose) may improve locoregional tumour control in non-small cell lung cancer (NSCLC) in comparison to conventional fractionation (5 fractions per week, 2 Gy single dose).

DETAILED DESCRIPTION:
This study is a randomized multicentric trial. Within this study an accelerated irradiation schedule (7 fractions per week, 2 Gy single dose) will be compared with the currently used conventional fractionation schedule (5 fractions per week, 2 Gy single dose) for postoperative radiotherapy with photons or protons in patients with NSCLC. The primary endpoint is locoregional tumour control after 36 months. Secondary endpoints are overall survival of patients, local recurrence-free and distant metastases-free survival after 36 months, acute and late toxicity as well as quality of life for both treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed non-small cell lung cancer
* previous tumor resection with curative intention
* postoperative indication for irradiation (> pN1 and/ or R1)
* R2-resection or recurrence postoperative/after adjuvant chemotherapy diagnosed by the restaging-imaging
* exclusion of distant metastases (M0)
* age > 18 years
* good general condition (ECOG performance status 0 or 1)
* written informed consent
* appropriate compliance to ensure close follow-up
* women of childbearing age: adequate contraception

Exclusion Criteria:

* histologically confirmed small cell lung cancer
* distant metastases
* no written informed consent or lack of cooperation relating to therapy or follow-up
* previous (< 5 years) or concomitant other malignant disease (exception: malignant disease, which is very likely healed and not influenced therapy or follow up of the non-small cell lung cancer, e.g. carcinoma in-situ, basaliomas, very early skin cancers)
* for proton therapy: heart pacemaker
* previous radiotherapy of the thorax or lower neck region
* pregnancy or lactation
* participation in another intervention study or not completed follow-up of a intervention study. Exceptions are psychological studies, supportive or observation studies, the previous therapy of non-small cell lung cancer is in accordance with the guideline and the participation in radiotherapy studies is not excluded in the trial protocol of the previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
assessment of local tumor control | 36 months after therapy
  Local tumor control will be assessed by appropriate non-invasive (CT or PET-CT) and if necessary invasive examination methods (bronchoscopy with biopsy).

SECONDARY OUTCOMES:
overall survival | 36 months after therapy
  Follow-up visits should be continued in all patients until death. Otherwise patients will be censored with date of the last follow-up.
local recurrence-free survival | 36 months after therapy
  Local-recurrences will be assessed by appropriate non-invasive (CT or PET-CT) and if necessary invasive examination methods (bronchoscopy with biopsy).
acute toxicity | Comparison after 20, 50, 100 and 200 patients have been treated. This number of patients is expected to be included after 6, 12, 18 and 40 months.
  The occurrence of acute side effects (up to 90 days after start of treatment) will be recorded and documented based on CTCAE 4.0.
quality of life | 36 months after therapy
  The assessment of quality of life is carried out using the established EORTC QLQ-C30 questionnaire and the additional lung module QLQ-LC13. Quality of life will be documented immediately before the start of therapy, after completion of postoperative radiotherapy and at every follow-up visit.
distant metastases-free survival | 36 months after therapy
  Distant metastases will be assessed by PET-CT or abdominal sonography and chest x-ray.
late toxicity | Comparison after 20, 50, 100 and 200 patients have been treated. This number of patients is expected to be included after 6, 12, 18 and 40 months.
  The occurrence of late side effects will be recorded and documented based on CTCAE 4.0 after every follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Bütof, Dr., Principal Investigator — Dresden University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology
Locations (9):
- Germany (8):
  - Universitätsklinikum Dresden, Department of Radiation Therapy and Radiation Oncology, Dresden
  - Universitätsklinikum Freiburg, Department of Radiation Therapy and Radiation Oncology, Freiburg im Breisgau
  - Praxis für Strahlentherapie Hamburg-Harburg, Hamburg
  - Universitätsklinikum des Saarlandes, Department of Radiotherapy and Radiation Oncology, Homburg
  - Klinikum der Universität München,Department of Radiation Therapy and Radiation Oncology, München
  - Klinikum rechts der Isar, Technische Universität München, Department of Radiation Therapy and Radiation Oncology, München
  - Marienhospital Stuttgart, Department of Radiotherapy and Palliative Medicine, Stuttgart
  - Universitätsklinikum Tübingen, Department of Radiation Therapy and Radiation Oncology, Tübingen
- SPZOZ MSW; Warmia & Mazury Oncology Center; Warmia & Mazury Medical University, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butof R, Koi L, Lock S, Appold S, Drewes S, Koschel D, Kotzerke J, Nestle U, Adebahr S, Zips D, Heinzelmann F, Hehr T, Bucher D, Heide J, Belka C, Manapov F, Wasilewska-Tesluk E, Fleckenstein J, Krause M, Troost EGC, Baumann M. Accelerated vs. conventionally fractionated postoperative radiotherapy of non-small cell lung cancer-final results of the prematurely terminated PORTAF trial. Strahlenther Onkol. 2025 Jul 15. doi: 10.1007/s00066-025-02422-y. Online ahead of print. PMID 40663146
- [Derived] Butof R, Simon M, Lock S, Troost EGC, Appold S, Krause M, Baumann M. PORTAF - postoperative radiotherapy of non-small cell lung cancer: accelerated versus conventional fractionation - study protocol for a randomized controlled trial. Trials. 2017 Dec 20;18(1):608. doi: 10.1186/s13063-017-2346-0. PMID 29262836